CLINICAL TRIAL: NCT06472362
Title: Deep-learning Derived Chest Computed Tomography (CT) Biomarkers as Prognostic Predictors in Systemic Sclerosis Associated Interstitial Lung Disease (SSc-ILD)
Brief Title: Chest CT Biomarkers as Prognostic Predictors in SSc-ILD
Status: Enrolling by invitation | Type: Observational
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Collaborators: Imperial College London (Other); Royal Free and University College Medical School (Other); The Leeds Teaching Hospitals NHS Trust (Other); Hannover Medical School (Other); University of Siena (Other); Università Politecnica delle Marche (Other); Azienda Ospedaliero Universitaria di Sassari (Other); Bichat Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RBH2
Record Dates: First submitted 2024-06-11; First posted 2024-06-25 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: HRCT biomarkers — HRCT imaging biomarkers of airways, vessels, and overall extent of fibrosis

SUMMARY:
The goal of this retrospective observational study is to investigate whether novel imaging biomarkers of airways, vessels, and overall extent of fibrosis at baseline predict ILD progression, vasculopathy development, and survival in SSc-ILD.

DETAILED DESCRIPTION:
Interstitial lung disease (ILD or lung fibrosis=stiffening of the lungs by scar tissue) develops in over half of patients with systemic sclerosis (SSc). Whilst ILD remains stable in some patients, at least a third have progressively increasing fibrosis. There is a pressing need for accurate indicators that identify a) patients at higher risk of progression, needing immediate treatment to prevent further irreversible ILD; and b) patients at lower risk, not needing treatment.

In this study the prognostic potential and accuracy of machine-learning derived biomarkers to evaluate abnormalities that are difficult to quantify visually will be investigated. Whether novel high resolution computed tomography (HRCT) imaging biomarkers of airways, vessels, and overall extent of fibrosis at baseline can predict ILD progression, vasculopathy development, and survival will be investigated in a cohort of approximately 1,000 SSc-ILD patients.

The algorithm scores will be evaluated against survival using Cox proportional hazards modelling, while mixed effects model analysis will be used to assess links with change in lung function: forced vital capacity (FVC), diffusing capacity for carbon monoxide (DLco), and carbon monoxide transfer coefficient (Kco). The airway algorithm measuring traction bronchiectasis (dilatation of the airways due to surrounding fibrosis) may predict worsening of FVC, reflective of ILD progression. The vessel algorithm may predict decline in KCO, a marker of pulmonary vascular involvement. Exploratory analyses evaluating change in HRCT fibrosis extent over time for patients with repeat HRCTs will also be performed, and whether composite outcomes of change in HRCT and lung function variables improve long term outcome prediction and pave the way to their use in clinical trials and routine clinical use. Patients with trivial changes on CT will also be included to assess for very early changes that could be predictive of future decline. These algorithms will be combined with the findings of our previous study, which suggest that a certain type of pattern on CT called UIP predicts shorter survival.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with SSc
* ≥18 years old
* HRCT between 01/01/1990 and 31/12/2019

Exclusion Criteria:

* Patients who do not have SSc
* <18 years old
* lack of availability of HRCT imaging data

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Secondary/tertiary care patients with SSc
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Survival | 15 years
  Transplant-free survival
Pulmonary hypertension | 15 years
  Development of pulmonary hypertension
Decline in FVC | 15 years
  Change in lung function measure FVC
Decline in DLCO | 15 years
  Change in lung function measure DLCO
Decline in KCO | 15 years
  Change in lung function measure KCO

CONTACTS AND LOCATIONS:
Overall Officials: Elisabetta A Renzoni, Principal Investigator — Royal Brompton and Harefield Hospitals
Locations (7):
- Bichat-Claude Bernard hospital, Paris, France
- Hanover Medical School, Hanover, Germany
- Italy (3):
  - Marche Polytechnic University, Ancona
  - Sassari University, Sassari
  - Siena University Hospital, Siena
- United Kingdom (2):
  - Leeds Hospital/University of Leeds, Leeds
  - Royal Brompton Hospital, London

IPD SHARING:
Plan to Share IPD: No